CLINICAL TRIAL: NCT07033910
Title: The Effect of Extracorporeal Sepsis Adsorption Column Use on Plasma Syndecan-1 Level and Mortality in Sepsis Patients
Brief Title: Effect of Sepsis Adsorption Column on Syndecan-1 and Mortality
Status: Completed | Type: Observational
Sponsor: Oral MENTEŞ (Other)
Responsible Party: Sponsor-Investigator, Oral MENTEŞ, Specialist Dr. Oral MENTEŞ (Chest Diseases and Intensive Care Specialist), Gulhane School of Medicine
Organization: Gulhane School of Medicine (Other)
Other Study IDs: GulhaneSM 2023/93; 001 (Other: Buy Pharma Ecza Deposu San. Tic. Ltd.)
Record Dates: First submitted 2025-04-25; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Sepsis; Syndecan 1; Extracorporeal Sepsis Adsorption Column
Keywords: Cytokine filter; intensive care unit; Interleukin-6; sepsis; sepsis adsorption column; Syndecan-1
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The remaining 8-10 mL venous blood samples from the routine blood collection of the patients included in the study were collected in red capped tubes. The blood samples were centrifuged at 4000 rpm for 10 minutes and serum was separated. The serum samples were stored in clean and dry ependorf tubes at -80°C until analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Adsorption Column Used: Consisted of 43 patients. Sepsis adsorption column used. After the initiation of fluid and antibiotic therapy according to the Surviving Sepsis Campaign 2021 Guidelines, an additional routine sepsis adsorption column (Biosky® MG350) was used within 48-72 hours. Clinical status, response to treatment, and plasma Syndecan-1 levels, among all laboratory variables, were evaluated within the first 24 hours following the filter application.
  Interventions: Device: sepsis adsorption column
- Standard Sepsis Treatment Only: Consisted of 48 patients. Sepsis adsorption column not used. Patients receiving only fluid and antibiotic therapy, with clinical status, treatment response, and plasma Syndecan-1 levels, along with other laboratory variables, evaluated within the 48-72 hour period.

INTERVENTIONS:
Device: sepsis adsorption column — after the initiation of fluid and antibiotic therapy according to the Surviving Sepsis Campaign 2021 Guidelines, an additional routine sepsis adsorption column (Biosky® MG350) was used within 48-72 hours.
  Groups: Adsorption Column Used

SUMMARY:
This observational, cross-sectional, single-center study aims to investigate the effect of extracorporeal sepsis adsorption column therapy on plasma Syndecan-1 levels and clinical outcomes in patients with sepsis. The study was conducted in the Internal Medicine Intensive Care Unit of Gülhane Training and Research Hospital. Patients were divided into two groups: one group received standard sepsis treatment along with an extracorporeal adsorption column (Biosky® MG350), while the other group received only standard treatment. Clinical and laboratory parameters, including Syndecan-1 levels, were evaluated to assess the potential impact of the adsorption column on sepsis-related outcomes.

DETAILED DESCRIPTION:
This single-center, cross-sectional, and observational study aims to evaluate the effect of extracorporeal sepsis adsorption column use on plasma Syndecan-1 levels and mortality in patients diagnosed with sepsis. The study was conducted in the Internal Medicine Intensive Care Unit of Gülhane Training and Research Hospital between May 25, 2023, and June 9, 2024.

Patients who met the inclusion criteria were divided into two groups:

Group 1: Patients received standard sepsis treatment, including fluid and antibiotic therapy according to the Surviving Sepsis Campaign 2021 Guidelines, in addition to extracorporeal sepsis adsorption column (Biosky® MG350) therapy applied within 48-72 hours of ICU admission.

Group 2: Patients received only fluid and antibiotic therapy, without the use of a sepsis adsorption column.

In both groups, plasma Syndecan-1 levels and various clinical and laboratory parameters were evaluated. These included APACHE II score, SOFA score, Charlson Comorbidity Index (CCI), comorbidities, infection focus, respiratory support status, vasopressor/inotrope requirement, laboratory values (including IL-6 and lactate), presence of acute kidney injury, need for hemodialysis, duration of ICU stay, and survival times.

The only treatment-related difference between the groups was the use of the adsorption column. Clinical and laboratory data were collected at standardized time intervals in each group to allow for comparison.

The study is designed to provide insight into whether the use of extracorporeal sepsis adsorption therapy has an observable impact on endothelial biomarkers such as Syndecan-1 and on patient outcomes in sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Patients (Patient or relative) who accepted and signed the informed consent form and approved participation in the study
* Patients over 18 years of age
* Patients diagnosed with sepsis/septic shock

Exclusion Criteria:

* The Informed Voluntary Consent Form has not been signed by him/herself and his/her legal heir
* Patients with sepsis who died within the first 24 hours after admission to the internal medicine intensive care unit and within the first 24 hours after sepsis diagnosis and within the first 24 hours after administration of sepsis adsorption column
* Patients in Group-1 who could not receive extracorporeal hemoperfusion for any reason or who could not be started and completed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gülhane Training and Research Hospital, Department of Internal Medicine Intensive Care Unit
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-06-09 (Actual); Study Completion 2024-06-09 (Actual)

PRIMARY OUTCOMES:
Plasma Syndecan-1 Level Following Sepsis Adsorption Column Treatment | Measured within 24 hours after cytokine adsorption column application in the adsorption column used group and at 48-72 hours after ICU admission in the standard sepsis treatment only group.
  Plasma Syndecan-1 levels (ng/mL) will be measured in patients diagnosed with sepsis. In the adsorption column used group, Syndecan-1 levels will be assessed within the first 24 hours following the administration of the extracorporeal sepsis adsorption column (Biosky® MG350), which is applied within 48-72 hours after ICU admission. In the standard sepsis treatment only group, Syndecan-1 levels will be measured at the 48-72 hour mark after ICU admission. The primary outcome is the comparison of Syndecan-1 levels between the two groups to evaluate the effect of the adsorption column on endothelial injury..

SECONDARY OUTCOMES:
Change in Serum Lactate Levels | From baseline (prior to adsorption column) to 24 hours after treatment in adsorption column used group; and from ICU admission to 48-72 hours in standard sepsis treatment only group.
  Comparison of median serum lactate levels (mmol/L) before and after treatment in both groups. The difference in lactate levels will be used to assess the metabolic response to treatment and organ perfusion improvement.
Post-Treatment Plasma Interleukin-6 (IL-6) Levels | At 24 hours post-treatment in adsorption column used group and 48-72 hours in standard sepsis treatment only group.
  Measurement of plasma IL-6 levels (pg/mL) to evaluate the inflammatory response in both groups.
Vasopressor/Inotrope Dose Correlation With Syndecan-1 Levels | At 24 hours post-treatment in adsorption column used group and 48-72 hours in standard sepsis treatment only group.
  Assessment of the correlation between plasma Syndecan-1 levels (ng/mL) and vasopressor/inotrope dose requirements (µg/kg/min).

CONTACTS AND LOCATIONS:
Overall Officials: HUSEYIN L YAMANEL, MD, PhD, Study Director — GULHANE SM
Locations (1):
- Gülhane Training and Research Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) generated from this study, including de-identified demographic, clinical, laboratory, and outcome data, will be made available upon reasonable request. Data sharing will be facilitated after publication of the primary results to support further research in sepsis biomarkers and treatment effects. Data requests can be submitted to the corresponding author, who will review proposals for scientific merit and ethical compliance before granting access. Data will be shared under a data use agreement to ensure confidentiality and proper use.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available for sharing starting 6 months after the publication of the primary study results and will remain available for a period of 5 years thereafter.
Access Criteria: De-identified participant data will be shared with researchers who submit a clear research plan. Data sharing requires approval by the study team and signing a data use agreement to protect privacy.

REFERENCES:
- [Background] Vivas MC, Villamarin Guerrero HF, Tascon AJ, Valderrama-Aguirre A. Plasma interleukin-6 levels correlate with survival in patients with bacterial sepsis and septic shock. Interv Med Appl Sci. 2021 Aug 2;11(4):224-230. doi: 10.1556/1646.2020.00006. eCollection 2021 Aug. PMID 36343289
- [Background] Hawchar F, Laszlo I, Oveges N, Trasy D, Ondrik Z, Molnar Z. Extracorporeal cytokine adsorption in septic shock: A proof of concept randomized, controlled pilot study. J Crit Care. 2019 Feb;49:172-178. doi: 10.1016/j.jcrc.2018.11.003. Epub 2018 Nov 10. PMID 30448517
- [Background] Becker S, Lang H, Vollmer Barbosa C, Tian Z, Melk A, Schmidt BMW. Efficacy of CytoSorb(R): a systematic review and meta-analysis. Crit Care. 2023 May 31;27(1):215. doi: 10.1186/s13054-023-04492-9. PMID 37259160
- [Background] Schadler D, Pausch C, Heise D, Meier-Hellmann A, Brederlau J, Weiler N, Marx G, Putensen C, Spies C, Jorres A, Quintel M, Engel C, Kellum JA, Kuhlmann MK. The effect of a novel extracorporeal cytokine hemoadsorption device on IL-6 elimination in septic patients: A randomized controlled trial. PLoS One. 2017 Oct 30;12(10):e0187015. doi: 10.1371/journal.pone.0187015. eCollection 2017. PMID 29084247
- [Background] Friesecke S, Stecher SS, Gross S, Felix SB, Nierhaus A. Extracorporeal cytokine elimination as rescue therapy in refractory septic shock: a prospective single-center study. J Artif Organs. 2017 Sep;20(3):252-259. doi: 10.1007/s10047-017-0967-4. Epub 2017 Jun 6. PMID 28589286
- [Background] Anand D, Ray S, Srivastava LM, Bhargava S. Evolution of serum hyaluronan and syndecan levels in prognosis of sepsis patients. Clin Biochem. 2016 Jul;49(10-11):768-76. doi: 10.1016/j.clinbiochem.2016.02.014. Epub 2016 Mar 4. PMID 26953518
- [Background] Lipowsky HH, Gao L, Lescanic A. Shedding of the endothelial glycocalyx in arterioles, capillaries, and venules and its effect on capillary hemodynamics during inflammation. Am J Physiol Heart Circ Physiol. 2011 Dec;301(6):H2235-45. doi: 10.1152/ajpheart.00803.2011. Epub 2011 Sep 16. PMID 21926341
- [Background] Gotte M. Syndecans in inflammation. FASEB J. 2003 Apr;17(6):575-91. doi: 10.1096/fj.02-0739rev. PMID 12665470
- [Background] Saunders S, Jalkanen M, O'Farrell S, Bernfield M. Molecular cloning of syndecan, an integral membrane proteoglycan. J Cell Biol. 1989 Apr;108(4):1547-56. doi: 10.1083/jcb.108.4.1547. PMID 2494194
- [Background] Liu Z, Meng Z, Li Y, Zhao J, Wu S, Gou S, Wu H. Prognostic accuracy of the serum lactate level, the SOFA score and the qSOFA score for mortality among adults with Sepsis. Scand J Trauma Resusc Emerg Med. 2019 Apr 30;27(1):51. doi: 10.1186/s13049-019-0609-3. PMID 31039813
- [Background] Nichol AD, Egi M, Pettila V, Bellomo R, French C, Hart G, Davies A, Stachowski E, Reade MC, Bailey M, Cooper DJ. Relative hyperlactatemia and hospital mortality in critically ill patients: a retrospective multi-centre study. Crit Care. 2010;14(1):R25. doi: 10.1186/cc8888. Epub 2010 Feb 24. PMID 20181242
- [Background] Garcia-Alvarez M, Marik P, Bellomo R. Sepsis-associated hyperlactatemia. Crit Care. 2014 Sep 9;18(5):503. doi: 10.1186/s13054-014-0503-3. PMID 25394679
- [Background] Faix JD. Biomarkers of sepsis. Crit Rev Clin Lab Sci. 2013 Jan-Feb;50(1):23-36. doi: 10.3109/10408363.2013.764490. PMID 23480440
- [Background] Ronco C, Chawla L, Husain-Syed F, Kellum JA. Rationale for sequential extracorporeal therapy (SET) in sepsis. Crit Care. 2023 Feb 7;27(1):50. doi: 10.1186/s13054-023-04310-2. PMID 36750878
- [Background] Hanasawa K. Extracorporeal treatment for septic patients: new adsorption technologies and their clinical application. Ther Apher. 2002 Aug;6(4):290-5. doi: 10.1046/j.1526-0968.2002.00449.x. PMID 12164799
- [Background] Jaber BL, Pereira BJ. Extracorporeal adsorbent-based strategies in sepsis. Am J Kidney Dis. 1997 Nov;30(5 Suppl 4):S44-56. doi: 10.1016/s0272-6386(97)90542-4. PMID 9372979
- [Background] David S, Bode C, Putensen C, Welte T, Stahl K; EXCHANGE study group. Adjuvant therapeutic plasma exchange in septic shock. Intensive Care Med. 2021 Mar;47(3):352-354. doi: 10.1007/s00134-020-06339-1. Epub 2021 Jan 20. No abstract available. PMID 33471132
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Piotti A, Novelli D, Meessen JMTA, Ferlicca D, Coppolecchia S, Marino A, Salati G, Savioli M, Grasselli G, Bellani G, Pesenti A, Masson S, Caironi P, Gattinoni L, Gobbi M, Fracasso C, Latini R; ALBIOS Investigators. Endothelial damage in septic shock patients as evidenced by circulating syndecan-1, sphingosine-1-phosphate and soluble VE-cadherin: a substudy of ALBIOS. Crit Care. 2021 Mar 19;25(1):113. doi: 10.1186/s13054-021-03545-1. PMID 33741039
- [Background] Dugar S, Choudhary C, Duggal A. Sepsis and septic shock: Guideline-based management. Cleve Clin J Med. 2020 Jan;87(1):53-64. doi: 10.3949/ccjm.87a.18143. Epub 2020 Jan 2. PMID 31990655
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- See also: Related Info — https://tez.yok.gov.tr/UlusalTezMerkezi/